CLINICAL TRIAL: NCT03543267
Title: Feasibility Study on Neurocognitive Plasticity in Patients With Focal and Drug-resistant Epilepsy, Before and After Surgery. Evaluation by Functional and Anatomic Neuroimaging
Brief Title: Study on Neurocognitive Plasticity in Patients With Focal and Drug-resistant Epilepsy
Acronym: FaisPLASTICITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC17.018
Record Dates: First submitted 2018-05-14; First posted 2018-06-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- epileptic Patients (Experimental)
  Interventions: Other: MRI exam

INTERVENTIONS:
Other: MRI exam — MRI before and after resection surgery

SUMMARY:
This study consist of define anatomo-functional reorganization (plasticity) profiles for the mentioned cognitive functions, before surgery (chronic plasticity induced by the epileptogenic zone) in patients with drug-resistant epilepsy.

For that, patients will have 2 MRI examinations, one before surgery and the second, between 3 and 8 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of pharmaco-resistant focal epilepsy
* Patient candidate for surgery to resect the epileptogenic zone
* Patients affiliated to a social security scheme or beneficiaries of such a scheme
* Patients with French as their mother tongue
* Patients who have given signed informed consent before performing any procedure related to the study.

Exclusion Criteria:

* Contraindication to performing an MRI:
* Intellectual disability objectified by a Mini Mental Score (MMS) score <24 in the year preceding inclusion,
* Existence of a severe condition in general: cardiac, respiratory, hematological, renal, hepatic, cancerous,
* Participation in other research protocols underway with exclusion period or in the previous week,
* Persons referred to in Articles L1121-5 to L1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
to define anatomo-functional reorganization (plasticity) profiles by functional MRI for the mentioned cognitive functions, before surgery (chronic plasticity induced by the epileptogenic zone) in patients with drug-resistant epilepsy. | One hour and thirty minutes
  The outcome measure is the hemispheric lateralization index (IL) before surgery measured by functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Monica BACIU, PhD, Principal Investigator — Centre National de la Recherche Scientifique, France
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France